CLINICAL TRIAL: NCT02409966
Title: Impact of Different Protocols for Treatment of Chronic Periodontitis on the Following Patient-centered Variables: Oral Health Related Quality of Life and Experiences of Fear, Anxiety and Pain: a 6 Month Randomized Clinical Trial
Brief Title: Effect of Periodontitis Treatment on Quality of Life and Experiences of Fear, Anxiety and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taubate (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 552264/2011-3; 521-10 (Other: Ethics committee); CAAE 07172212.3.0000.514 (Other: Ethics committee)
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Periodontitis
Keywords: periodontitis; therapeutics; quality of life; fear; anxiety; pain
MeSH Terms: conditions — Periodontitis; Anxiety Disorders; Pain | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quadrant-wise scaling (Active Comparator): Patients underwent quadrant scaling under local anesthesia in four weekly sections.
  Interventions: Procedure: Quadrant-wise scaling
- Full-mouth 24-hour scaling (Experimental): Patients underwent full-mouth scaling under local anesthesia in two sections within 24 hours.
  Interventions: Procedure: Full-mouth 24-hour scaling

INTERVENTIONS:
Procedure: Quadrant-wise scaling — Patients underwent quadrant scaling under local anesthesia in four weekly sections. Three experienced trained periodontists carried out debridement procedures of both protocols with manual Gracey and McCall curettes and Hirschfield files.
  Oral hygiene instructions were given for all participants and oral supplies were provided for the duration of the study.
  Arms: Quadrant-wise scaling
Procedure: Full-mouth 24-hour scaling — Patients underwent full-mouth scaling under local anesthesia in two sections within 24 hours. Three experienced trained periodontists carried out debridement procedures of both protocols with manual Gracey and McCall curettes and Hirschfield files.
  Oral hygiene instructions were given for all participants and oral supplies were provided for the duration of the study.
  Arms: Full-mouth 24-hour scaling

SUMMARY:
There are different protocols to treat gum diseases. One relevant differential aspect is related to time. There are protocols that usually takes one to two months to be completed while other are completed within 24 hours. Although both protocols seem to provide clinically similar improvements, there are some positive aspects related to the short-term one. Among them lower number of clinical sessions, easier schedule and costs advantages. However, there are many other relevant aspects that can be helpful for patients and clinicians decisions regarding type of treatment.

This study evaluates if and how clinically effective protocols used to treat periodontitis affect quality of life related to individual's oral statuses. In addition, the experiences of fear, anxiety and pain before and after these specific protocols are monitored.

DETAILED DESCRIPTION:
Most randomized controlled clinical trials regarding the effects of non-surgical periodontal treatment have focused on objective parameters. Their effects on patient-centered variables have been received very little attention. After determining clinical therapeutic efficacy, this study compared over 6 months the effects of two different forms of non-surgical periodontal therapy - scaling and root planing per quadrant (SRP) and one-stage full-mouth disinfection (FMD) - on scores of quality of life, fear, anxiety and pain of moderate chronic periodontitis. Initially, the sample size was calculated considering protocols' clinical efficacy. Specifically for the present study it was verified if the initial sample size would be enough for analysis of the subjective variables.

Patients registered in dental care centers from University of Taubate, Taubate - Sao Paulo, Brazil and Federal University of Minas Gerais, Belo Horizonte - Minas Gerais, Brazil were informed about the objectives and methods of the study, being consecutively included in the study only after signing an informed consent form. Selected participants were randomly allocated to one of the treatment groups by a closed envelope system. According to the designated group, participants receive either conventional quadrant scaling in four weekly sections or full-mouth scaling within 24 hours.

Two experienced trained periodontists carried out debridement procedures of both protocols with manual Gracey and McCall curettes and Hirschfield files.

Specific validated instruments were used to evaluate subjective variables. Oral Impacts on Daily Performance (OIDP) and Oral Health and Quality of Life (OHQoL-UK) measured quality of life while Dental Fear Survey (DFS), Dental Anxiety Scale (DAS) questionnaires and, Visual Analog Scale (VAS) measured experienced fear, anxiety and pain, respectively.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate chronic periodontitis
* smokers or non-smokers
* at least 18 natural teeth

Exclusion Criteria:

* regular use or use in the previous 3 months of antibiotics or anti-inflammatory drugs
* regular use (twice a day) of mouthwashes
* sensitivity or allergy to oral hygiene products
* patients undergoing periodontal therapy including dental scaling and root planing procedures in the 12 months preceding the start of the study
* bifurcation or trifurcation class III lesions
* the need for antibiotic prophylaxis for periodontal clinical examination/treatment
* removable partial dentures, fixed or removable orthodontic devices
* pregnancy and lactation
* medical or psychological disorder that could affect the ability of the questionnaires' understanding

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Oral health related quality of life | changes in OIDP and OHQoL scores from baseline to 6 months
Scale of self-reported pain | changes in VAS scores from baseline to 1 month
Fear and anxiety | changes in DFS and DAS scores from baseline to 6 months

OTHER OUTCOMES:
Periodontal pocket depth (mm) and clinical attachment level (mm) were measure at baseline and at 6 months after active periodontal treatment. | from baseline to 6 months